CLINICAL TRIAL: NCT00458146
Title: A Phase 2, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of 60mg of MM-093 Versus Placebo in Patients With Active Rheumatoid Arthritis on Stable Doses of Methotrexate
Brief Title: A Phase 2 Study to Evaluate the Efficacy and Safety of 60mg of MM-093 in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Responsible Party: Merrimack Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MM-093-01-201
Record Dates: First submitted 2007-04-05; First posted 2007-04-09 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): MM-093
  Interventions: Drug: MM-093
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: MM-093

INTERVENTIONS:
Drug: MM-093 — 60mg MM-093/week as a subcutaneous injection for 3 months

SUMMARY:
The purpose of this study is to determine whether MM-093 is safe and effective in the treatment of RA.

DETAILED DESCRIPTION:
To evaluate the safety and tolerability of 60 mg of MM-093 in patients who have active RA despite MTX background therapy.

ELIGIBILITY:
Inclusion Criteria:

* Meet American College of Rheumatology (ACR) criteria for RA.
* Have active RA consisting of > or equal to 6 tender joints and > or equal to 6 swollen joints and one of the following:CRP or ESR levels of ULN
* Have an ACR functional class of I-III.
* Have had RA for at least 6 months.
* Had disease onset at > 16 years of age.
* Aged 18 - 80 years.
* Currently being treated with a stable, well tolerated weekly dose of MTX between 10-25 mg for at least 6 consecutive prior to screening visit.
* Currently being treated with folic/folinic acid in conjunction with their MTX treatment.

(Note: Patients may begin folic/folinic acid treatment after their screening visit, but must remain on stable dose for two weeks before undergoing the Day 1 assessments.)

* Willing to remain on a constant, weekly dose of MTX and folic/folinic acid through out the duration of the study.
* Understand, sign, and date the written, voluntary informed consent form at the screening visit prior to any protocol - specific procedures being performed.
* Be able and willing to comply with study visits and procedures per protocol.
* Women of childbearing potential must use a medically acceptable means of birth control in an effective manner and agree to continue its use during the study and for 4 weeks after the last dose of study drug. Women who have had a complete surgical hysterectomy or are postmenopausal (absence of menstrual period for at least one year or > 52 years old) are exempt from this requirement. Medically acceptable forms of birth control include oral contraceptives, injectable or implantable methods, intrauterine devices, tubal ligation (if performed more than 1 year before screening), or properly used barrier contraception. Additionally, the use of condoms is suggested as an adjunct to the methods previously addressed to protect against sexually transmitted diseases and to provide additional protection against accidental pregnancy.
* Sexually active men must agree to use a medically acceptable form of contraception during the study and continue for 4 weeks after the last dose of study drug.
* Able to store patient kit/cooler containing drug in a refrigerator at home.

Exclusion Criteria:

* Patient will be excluded if any of the following prior medications are currently being used or have used within the designated time interval before the screening visit:

  1. Any B - cell or antibody depleting therapy , including plasmaphoresis or Prosorba columns (6 months)
  2. Leflunomide, Adalimumab (Humira)(3 months)
  3. Investigational biologics (2 months)
  4. Infliximab (Remicade) (2 months)
  5. Cyclosporine, sulphasalazine, auranofin, intramuscular gold, azathioprine, D-penicillamine, tacrolimus (6 weeks)
  6. Investigational small molecules (e.g. NSAIDS or Cox-2 inhibitors)(4 weeks)
  7. Use more than 10mg/day of prednisone or equivalent (4 weeks)
  8. Bolus intramuscular/intravenous (IM/IV) treatment with corticosteroids (>20 mg prednisone or equivalent)(4 weeks)
  9. Intra-articular corticosteroid injection (4 weeks)
  10. Etanercept (Enbrel) (4 weeks)
  11. Anakinra (Kineret) (2 weeks)
  12. Use of more than one NSAID (current)
  13. Dose of NSAID greater than maximum recommended dose in the product information (current)
* Significant concurrent medical diseases including:

  1. Cancer, or a history of cancer (other than successfully resected cutaneous basal and squamous cell carcinoma) within 5 years before the screening visit.
  2. Any condition for which participation in this study is judged by the physician to be detrimental to the patient, such as history of significant or unstable cardiac, pulmonary, gastrointestinal, neurological, or psychiatric disease, or a DMARD-related severe, potentially life threatening AE.
  3. Significant ongoing infection requiring systemic antibiotic, antifungal, antiviral, or anti-myobacterial therapy.
* Autoimmune or connective tissue disorder other than rheumatoid arthritis (e.g. Systemic Lupus Erythematosis, Scleroderma, or Psoriatic Arthritis)
* Grade 2 or above leukopenia (i.e. white blood cells < 3000/mm^3 [SI units: < 3.0 x 10^9/L)
* Thrombocytopenia or thrombocytosis (platelets > 125,000/mm^3 or > 1,000,000/mm^3 [SI units: < 125 x 10^9/L or > 1,000 x 10^9/L]), respectively.
* Grade 2 or above liver function abnormality(i.e. total bilirubin .1.5 x the upper limit of normal; or aspartate aminotransfersate [AST/SGOT] or alanine aminotransferase [ALT/SGPT]> 2.5 x upper limit of normal.
* Renal disease (including serum creatinine level > 1.5 x the upper limit of normal).
* Any history of immunodeficiency syndromes or infection with human immunodeficiency virus (HIV), or a history of hepatitis C or chronic hepatitis B.
* Pregnant or breastfeeding women or women planning to become pregnant during the study or within 4 weeks after the last dose of study drug.
* Any major surgery, including joint surgery, within 3 months before the screening visit.
* Scheduled elective surgery during the study participation.
* Participated in any previous clinical trial using MM-093 or have any prior exposure to MM-093.
* History of severe hypersensitivity to goat, sheep, or cow milk. (Patients who are lactose intolerant are not excluded).
* Any other condition that the investigator feels would jeopardize the integrity of the study (e.g. a CTCAE grade 2 or above clinical finding or laboratory result).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-02

PRIMARY OUTCOMES:
Evaluate the efficacy of MM-093 using ACR20 response rate | After three months of treatment

SECONDARY OUTCOMES:
Evaluate the efficacy of MM-093 using DAS-28 and EULAR | After three months of treatment

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Montgomery Rheumatology Associates, Montgomery, Alabama
  - East Valley Rheumatology & Osteoporosis, Gilbert, Arizona
  - Radiant Research, Scottsdale, Arizona
  - Arthritis Medical Center of the Central Coast, Santa Maria, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Denver Arthritis Clinic, Denver, Colorado
  - New England Research Associates, Trumbull, Connecticut
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - Paddock Park Clinical Research, Ocala, Florida
  - Arthritis Research of Florida, Inc., Palm Harbor, Florida
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Illinois Bone & Joint Institute, Morton Grove, Illinois
  - Wichita Clinic, Wichita, Kansas
  - Arthritis Center of Nebraska, Lincoln, Nebraska
  - Arthritis Center of Reno, Reno, Nevada
  - Arthritis Center and Carolina Bone and Joint, Charlotte, North Carolina
  - East Pennsylvania Rheumatology Association, Bethlehem, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Rheumatology and Internal Medicine, Amarillo, Texas
  - University of Utah Division of Rheumatology, Salt Lake City, Utah